CLINICAL TRIAL: NCT05531981
Title: Clinical Value of Minimal Residual Disease Detection Based on Human Papillomavirus Circulating Tumor DNA (HPV ctDNA) in Cervical Cancer
Brief Title: Detection of Minimal Residual Disease Based on HPV ctDNA in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); Peking University Cancer Hospital & Institute (Other); Precision Scientific (Beijing) Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: CC-MRD-1
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-08

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- initial surgical treatment group: After the patients were enrolled in the study according to the criteria, they were given standard treatment. The patients were followed up every 3~6 months within 2 years after treatment and every 6~12 months from 3 to 5 years after treatment, including general and gynecological physical examination, cervical or vaginal cytology test, HPV typing test, SCC, CA125, and imaging examination such as CT or MRI if necessary.
  Peripheral blood samples were collected to detect HPV E7 ctDNA before treatment, 2 weeks after surgery, (1 month after adjuvent radiotherapy if available) and at 6, 12, 18, 24, 30, and 36 months of follow-up.
  Interventions: Other: detect HPV E7 ctDNA
- initial concurrent chemoradiotherapy group: After the patients were enrolled in the study according to the criteria, they were given standard treatment. The patients were followed up every 3~6 months within 2 years after treatment and every 6~12 months from 3 to 5 years after treatment, including general and gynecological physical examination, cervical or vaginal cytology test, HPV typing test, SCC, CA125, and imaging examination such as CT or MRI if necessary.
  Peripheral blood samples were collected to detect HPV E7 ctDNA before treatment, 1 month after radiotherapy and at 6, 12, 18, 24, 30, and 36 months of follow-up.
  Interventions: Other: detect HPV E7 ctDNA

INTERVENTIONS:
Other: detect HPV E7 ctDNA — Peripheral blood was collected from the patients, and the copy number of HPV E7 gene in ctDNA was accurately detected by ddPCR

SUMMARY:
In this study, a large-scale cohort of cervical cancer patients was established in multiple centers. Minimal residual disease(MRD) was assessed by ddPCR detection of HPV E7 gene ctDNA to assess tumor burden and predict the risk of disease recurrence, so as to provide new biomarkers for precise treatment of cervical cancer patients. The study continued until 36 months after the end of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to assess MRD by detecting HPV E7 gene ctDNA to assess tumor burden and predict the risk of disease recurrence. According to the treatment methods, the patients were divided into two groups :(1) initial surgical treatment group (2) initial concurrent chemoradiotherapy group.

After the patients were enrolled in the study according to the criteria, they were given standard treatment. The patients were followed up every 3~6 months within 2 years after treatment and every 6~12 months from 3 to 5 years after treatment, including general and gynecological physical examination, cervical or vaginal cytology test, HPV typing test, SCC, CA125, and imaging examination such as CT or MRI if necessary.

Peripheral blood samples were collected to detect HPV E7 ctDNA before treatment, after treatment, and at 6, 12, 18, 24, 30, and 36 months of follow-up.

The primary endpoint is Disease-free survival (DFS, time from the treatment initiation to disease progression). Secondary endpoints include HPV ctDNA state before treatment, dynamic change trend of HPV ctDNA after treatment and overall survival (OS, time from the treatment initiation to death).

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis: cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma
* FIGO stage: IA2-IVA
* HPV typing: type 16 or 18
* ECOG 2-0
* The initial treatment was surgery (Cohort A) / concurrent chemoradiotherapy (Cohort B)

Exclusion Criteria:

* The diagnosis of cervical cancer was made within 3 years of other malignancies
* Pregnant or lactating women
* Refused to sign a consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A: Patients with cervical cancer who were initially treated with surgery in Peking Union Medical College Hospital, Peking University Cancer Hospital and Beijing Obstetrics and Gynecology Hospital, capital Medical University were enrolled in this study.
  Cohort B: Patients who were initially treated with concurrent chemoradiotherapy in Peking Union Medical College Hospital, Peking University Cancer Hospital and Beijing Obstetrics and Gynecology Hospital, capital Medical University were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | up to three years
  time from the treatment initiation to disease progression

SECONDARY OUTCOMES:
HPV ctDNA state before treatment | up to three years
  Peripheral blood was collected from the patients before treatment (surgery or chemotherapy), and the copy number of HPV E7 gene in ctDNA was accurately detected by ddPCR
Dynamic change trend of HPV ctDNA after treatment | up to three years
  Peripheral blood was collected from the patients after treatment ((2 weeks after surgery), 1 month after radiotherapy and at 6, 12, 18, 24, 30, and 36 months of follow-up), and the copy number of HPV E7 gene in ctDNA was accurately detected by ddPCR
Overall Survival | up to three years
  time from the treatment initiation to death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No